CLINICAL TRIAL: NCT06512441
Title: Vitamin B6 Assists in the Treatment of Inflammatory Bowel Disease
Brief Title: Vitamin B6 Aids in Treating Inflammatory Bowel Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, professor, Changhai Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VitB6
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Inflammatory Bowel Diseases
Keywords: VitaminB6; treatment
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Vitamin B 6; Therapeutics

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blind randomized controlled trial involving patients and healthcare providers
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental：VitaminB6 group (Experimental): Based on the standard treatment，VitaminB6 （10mg/tablet）is given orally once a day,one tablet each time,for 3 weeks.
  Interventions: Drug: Vitamin B6 Tablets; Drug: Placebo
- Placebo Comparator:Control group (Placebo Comparator): Based on the standard treatment，the same type of placebo tablets are given orally once a day,one tablet each time,for 3 weeks.
  Interventions: Drug: Vitamin B6 Tablets; Drug: Placebo

INTERVENTIONS:
Drug: Vitamin B6 Tablets — The experimental group was given a Vitamin B6 tablet（10mg/tablet）once a day for 3weeks, besides of the standard IBD treatment.
  Other Names: Treatment
Drug: Placebo — The control group was given a placebo tablet on the same type once a day for 3weeks, besides of the standard IBD treatment.
  Other Names: Control

SUMMARY:
Patients with IBD are randomized to oral administration of VitaminB6 and placebo based on the standard treatment, exploring whether VitaminB6 can increasee the clinical remission rateand improve the treatment effect of IBD patients.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a group of chronic idiopathic inflammatory intestinal diseases, mainly including ulcerative colitis and Crohn's disease, with increasing incidence in China and worldwide. The disease currently lacks a cure, with many patients experiencing relapses and requiring surgery, and an increased risk of cancer. There is substantial evidence suggesting a close relationship between body vitamin B6 levels and IBD.Thus,we design this clinical trial that aims to explore whether VitaminB6 can increasee the clinical remission rateand improve the treatment effect.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with IBD according to the consensus on the diagnosis and treatment of inflammatory bowel disease (Beijing, 2018, DOI: 10.19538/j.nk2018090106);
* Have complete medical history data;
* Volunteer to participate in this clinical trial and sign the informed consent form.

Exclusion Criteria:

* Patients with peripheral neuropathy;
* Patients with abdominal abscess, toxic megacolon, fulminant colitis, partial colectomy, or total colectomy;
* Patients with other autoimmune diseases, hematologic disorders, tumors, acute infections, severe liver or kidney dysfunction, severe conditions such as severe anemia, neutropenia, heart failure, organic heart disease, hepatitis B, cirrhosis, kidney disease, and psychiatric disorders;
* Patients who have taken vitamin B6 tablets in the past 3 months;
* Patients with a history of substance abuse;
* Pregnant or lactating women, or those planning to become pregnant within the next 6 months;
* Neurological disorders such as Alzheimer's disease, stroke, Parkinson's disease;
* Participation in other clinical trials in the past 6 months;
* Incomplete medical records (including gender, age, diagnosis, colonoscopy results, pathological diagnosis results, and other demographic data);
* Currently taking: levodopa, phenobarbital, phenytoin sodium.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Clinical remission rate | Through study completion, an average of 6 months .
  To evaluate the improvement effect of clinical remission rate (Mayo score ≤ 2 points and no single sub-score>1 point; CDAl score<150) in IBD patients after 3 weeks of oral Vitamin B6 while taking routine treatment.

SECONDARY OUTCOMES:
Disease activity score of IBD patients | Through study completion, an average of 6 months .
  Modified Mayo score or CDAl score
Histological remission | Through study completion, an average of 6 months .
  Based on the Geboes scale. No or slight increase of chronic inflammatory infiltration in lamina propria, no neutrophils in lamina propria or epithelium, no persistent clinicai response of erosion, ulcer or granulation tissue.
Clinical response | Through study completion, an average of 6 months .
  Modified Mayo score decreased by 2 points and 30% from baseline+rectal bleeding score decreased by 1 point or absolute rectal bleeding score decreased by 1 point.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoshen Li, Principal Investigator — The First Affiliated Hospital of Naval Medical University; Shu Zhu, Study Director — The University of Science and Technology of China
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China